CLINICAL TRIAL: NCT05102890
Title: ESOGER PC: Implementation of a Socio-geriatric Telemedicine Tool in Primary Care to Support Needs Assessment for Older Adults
Brief Title: Implementation of a Telemedicine Tool in Primary Care for Older Adults
Acronym: ESOGER-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MP-02-2022-10160; 2022-IMPV-309559 (Other Grant/Funding Number: FRQS)
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Telemedicine tool as a pre-consultation assessment for older patients in the primary care setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients 65 years old and older will receive a pre-consultation screening questionnaire by phone prior to their virtual or in-person visit. A summary report based on the results of the questionnaire will be placed in the patient electronic chart for use by the clinician at the time of visit.
  Interventions: Other: ESOGER
- Control Group (No Intervention): Usual care in the primary care clinic

INTERVENTIONS:
Other: ESOGER — For patients in the intervention group, ESOGER will be administered by phone by a member of the clinic team prior to their virtual or in-persons consultation with their primary care provider. ESOGER is already available on an online platform for data entry. Based on feedback our team obtained from interviews with current users of ESOGER, administration of the tool is expected to take between 5 and 10 minutes. A report summarizing the health and social status of the patient along with flagged potential vulnerabilities will be generated automatically by the online ESOGER platform. This report will then be uploaded to the patient's electronic chart by a member of the clinic and made available for the primary care provider at the time of the consultation.
  Arms: Intervention group

SUMMARY:
The pandemic has served a major catalyst propelling telehealth to the frontline of health care. For older adults who often live many chronic health problems, telehealth, which means to give medical check-ups by phone, email or by video conferencing, has become a lifeline to accessing a doctor when they need one. Even without the pandemic, telehealth can help ease access to care, especially for those living in rural areas who often need to travel long distances to see a doctor. However, there is a lack of telehealth tools that have been adapted for older patients. For example, only a few studies have looked at how well they work in improving outcomes for older patients like their quality of life, autonomy and use of health services. Telehealth could also lead to unfair differences between urban and rural patients who don't have the same access to technology. All these factors can make it difficult for family doctors to feel confident about using telehealth for their older patients. With telehealth likely to become mainstream for family doctors and older patients even after the pandemic, it is important to support the growing use of telehealth through tools that are adapted for older patients, fair and based on reliable evidence. This project aims to support the shift to telehealth in caring for older people living in the community by implementing and evaluating ESOGER, a telehealth support tool, in family medicine clinics. The ESOGER tool provides s a quick and reliable evaluation of the health and social needs of older patients. It can be done by phone making it accessible for everyone. This tool is expected to give family doctors a standardized and feasible way to determine the health and social needs of their older patients using telehealth which will help improve patients' autonomy, quality of life and health service use. The tool will be tested in four clinics in both urban and rural regions of Quebec to find out if it helped doctors better address their patients' needs and helped patients to live well at home. The study investigators will also study any differences in improvement between urban and rural older patients. They will discuss the results with the clinics and patient-partners to learn from their experiences and make the telehealth tool and the way to use it be as optimal as possible for family doctors to help maintain the health, quality of life and autonomy of older patients living at home.

DETAILED DESCRIPTION:
The goal of this project is to provide a readily-available solution to support an evidence-based shift to telemedicine in primary care by implementing and evaluating ESOGER as a pre-consultation telemedicine tool for older adults. Specifically, the objective of this project is to implement and evaluate the effectiveness of the ESOGER telemedicine tool in improving patient outcomes in rural and urban older patients. The effectiveness of the tool will be determined through a pilot randomized controlled trial in four university-affiliated interprofessional primary care clinics in the province of Quebec, Canada. Specifically, a 3-month pragmatic, multi-center, individually randomized, open-label and parallel-group trial design will be used. This design will evaluate the effectiveness of the tool under real-world conditions, allowing for site-specific adaptations to its implementation based on their needs and resources and producing results that can be generalized in routine practice settings. A 1:1 randomization ratio will be used to randomize patients to either receive the ESOGER tool or receive usual care. Participants will consist of those 65 years old and older with an upcoming virtual or in-person visit at one of the participating clinics who have consented to participate. A total of 480 participants expected to be recruited over the 3-month period. Baseline data on sociodemographic characteristics, self-reported quality of life and prior health service utilization will be collected by phone using an online questionnaire for patients in both study groups. The primary endpoint will consist of the EQ-5D score at the 3-month follow-up. The EQ-5D is a widely-used and validated 5-item patient-reported outcome measures (PROMS) tool that reflects patients' current perspective of their health, autonomy and quality of life. The EQ-5D index lies on a continuum from worst to best health, ranging from less than 0 to 1. Secondary endpoints will be unplanned health service use since the previous assessment (in last 3 months). An intention-to-treat analysis will be carried out for all study outcomes. A mixed effect model will be used to estimate the association between the use of ESOGER and outcomes accounting for the clustering of patients within study sites. A two-way interaction between the intervention group (ESOGER vs control group) and rural status (urban vs rural) will be included in the model to examine differences in impact for urban and rural older patients and potential areas of inequity. Analyses and interpretations will be carried out in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and older
* Patient of the participating primary care clinic with upcoming virtual or in-person primary care visit

Exclusion Criteria:

* unable to provide informed consent in English or French

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 452 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of life score at 3 months | The EQ-5D will be measured at study entry (time 0) and at study follow-up (3 months) for both the intervention and control group.
  The Euro-Qol 5D (EQ-5D), a highly validated quality of life questionnaire, will be used to measure the primary outcome. The EQ-5D score ranges from 0 (indicating worst health) to 1 (best health). The change in quality of life score will be measured as the difference in the EQ-5D score at 3 months minus the EQ-5D score at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Sourial, PhD, Principal Investigator — Université de Montréal
Locations (1):
- School of Public Health, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No